CLINICAL TRIAL: NCT02149199
Title: A Clinical Study Comparing Symbicort® 'as Needed' With Terbutaline 'as Needed' and With Pulmicort® Twice Daily Plus Terbutaline 'as Needed' in Adult and Adolescent Patients With Asthma.
Brief Title: A Clinical Study to Evaluate Symbicort Turbuhaler Used 'as Needed' in Adults and Adolescents With Asthma.
Acronym: SYGMA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D589SC00001; 2013-004474-96 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Symbicort "as needed"+placebo Pulmicort bid (Experimental): Symbicort (budesonide/formoterol) Turbuhaler 160/4.5 μg 'as needed' + Placebo Pulmicort Turbuhaler 200 μg bid
  Interventions: Drug: budesonide/formoterol 'as needed' + budesonide placebo bid
- terbutaline "as needed"+placebo Pulmicort bid (Active Comparator): terbutaline Turbuhaler 0.4 mg 'as needed' + placebo Pulmicort 200 μg Turbuhaler bid
  Interventions: Drug: terbutaline 'as needed' + placebo budesonide bid
- Pulmicort bid + terbutaline "as needed" (Active Comparator): Pulmicort 200 μg Turbuhaler bid + terbutaline 0.4 mg Turbuhaler 'as needed'
  Interventions: Drug: budesonide bid + terbutaline 'as needed'

INTERVENTIONS:
Drug: budesonide/formoterol 'as needed' + budesonide placebo bid — Symbicort (budesonide/ formoterol) 160/4.5 μg powder for inhalation 'as needed' plus Pulmicort placebo 200 μg powder for inhalation, 1 inhalation twice daily (morning and evening), 52-week treatment
  Arms: Symbicort "as needed"+placebo Pulmicort bid
Drug: terbutaline 'as needed' + placebo budesonide bid — Terbutaline 0.4 mg powder for inhalation 'as needed' plus placebo Pulmicort (budesonide) 200 μg powder for inhalation, 1 inhalation twice daily (morning and evening), 52-week treatment
  Arms: terbutaline "as needed"+placebo Pulmicort bid
Drug: budesonide bid + terbutaline 'as needed' — Pulmicort (budesonide) 200 μg powder for inhalation, 1 inhalation twice daily (morning and evening) plus terbutaline 0.4 mg powder for inhalation 'as needed', 52-week treatment
  Arms: Pulmicort bid + terbutaline "as needed"

SUMMARY:
The purpose of this study is to test if Symbicort® (budesonide/formoterol) Turbuhaler® is effective in treating asthma when used 'as needed' in patients with milder asthma. The efficacy of Symbicort® 'as needed' will be compared with: 1) terbutaline Turbuhaler® 'as needed' and with 2) Pulmicort (budesonide) Turbuhaler® twice daily plus terbutaline Turbuhaler® 'as needed'.

DETAILED DESCRIPTION:
A 52-week, double-blind, randomised, multi-centre, parallel-group, Phase III study in patients 12 years and older with asthma, evaluating the efficacy and safety of Symbicort® (budesonide/formoterol) Turbuhaler® 160/4.5 μg 'as needed' compared with terbutaline Turbuhaler® 0.4 mg 'as needed' and with Pulmicort® (budesonide) Turbuhaler® 200 μg twice daily plus terbutaline Turbuhaler® 0.4 mg 'as needed'

ELIGIBILITY:
INCLUSION CRITERIA 1. Provision of informed consent prior to any study specific procedures. For patients under-age, signed informed consent from both the patient and the patient's parent/legal guardian is required 2. Male or Female, ≥12 years of age 3. Documented diagnosis of asthma for at least 6 months prior to Visit 1 4. Patients who are in need of Step 2 treatment according to Global Initiative for Asthma guidelines 5. Patients treated with 'as needed' inhaled short-acting bronchodilator(s) only should have pre-bronchodilator Forced Expiratory Volume in one second (FEV1) ≥ 60 % of Predicted Normal (PN) and post-bronchodilator FEV1 ≥ 80 % PN 6. Patients treated with low stable dose of inhaled corticosteroid or leukotriene antagonist in addition to 'as needed' use of inhaled short-acting bronchodilator(s) should have pre-bronchodilator FEV1 ≥80 % PN 7. Patients should have reversible airway obstruction 8. To be randomized patients must have used Bricanyl Turbuhaler 'as needed' on at least 3 separate days during the last week of the run in period. EXCLUSION CRITERIA 1. Patient has a history of life-threatening asthma including intubation and intensive care unit admission 2. Patient has had an asthma worsening requiring change in treatment other than inhaled short-acting bronchodilator(s) within 30 days prior to Visit 1 or between Visits 1 and 2; or a treatment other than Bricanyl Turbuhaler from Visit 2 until randomization 3. Patient has required treatment with oral, rectal or parenteral glucocorticosteroids (GCS) within 30 days and/or depot parenteral GCS within 12 weeks prior to Visit 1 4. Smoker (current or previous) with a smoking history of ≥ 10 pack years 5. Pregnancy, breast-feeding or planned pregnancy during the study.

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3850 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M O'Byrne, MB, FRCP(C), FRSC, Principal Investigator — McMaster University, Hamilton, Canada
Locations (172):
- Australia (5):
  - Research Site, Bedford Park
  - Research Site, Concord
  - Research Site, Maroubra
  - Research Site, Murdoch
  - Research Site, Wollongong
- Brazil (7):
  - Research Site, Alphaville
  - Research Site, Botucatu
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (13):
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Plovdiv
  - Research Site, Razgrad
  - Research Site, Roman
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Velingrad
  - Research Site, Vratsa
- Canada (28):
  - Research Site, Edmonton, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Maple Ridge, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Cornwall, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kanata, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Victoriaville, Quebec
- Chile (3):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talcahuano
- China (14):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hohhot
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xuzhou
- Hungary (12):
  - Research Site, Balassagyarmat
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Hajdúnánás
  - Research Site, Mátészalka
  - Research Site, Miskolc
  - Research Site, Monor
  - Research Site, Nyírbátor
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
- Mexico (6):
  - Research Site, D.F.
  - Research Site, Durango
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Villahermosa
- Peru (4):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Piura
  - Research Site, Surco
- Philippines (4):
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (17):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Grudziądz
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Strzelce Opolskie
  - Research Site, Szczecin
  - Research Site, Słupca
  - Research Site, Tarnów
  - Research Site, Trzebnica
  - Research Site, Turek
  - Research Site, Zabrze
- Romania (6):
  - Research Site, Bragadiru
  - Research Site, Brasov
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Piteşti
  - Research Site, Timișoara
- Russia (22):
  - Research Site, Chelyabinsk
  - Research Site, Gatchina
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Petrozavodsk
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ulyanovsk
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Africa (7):
  - Research Site, Boksburg North
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, KwaDukuza
  - Research Site, Middelburg
  - Research Site, Queenswood
  - Research Site, Verulam
- South Korea (4):
  - Research Site, Bucheon-si
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Seoul
- Ukraine (10):
  - Research Site, Cherkasy
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- United Kingdom (5):
  - Research Site, Bath
  - Research Site, Coventry
  - Research Site, Mortimer Reading
  - Research Site, Royal Leamington Spa
  - Research Site, Trowbridge
- Vietnam (5):
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Đông Nãi

REFERENCES:
- [Derived] FitzGerald JM, O'Byrne PM, Bateman ED, Barnes PJ, Zheng J, Ivanov S, Lamarca R, Larsdotter U, Emerath U, Jansen G, Puu M, Alagappan VKT, Surmont F, Reddel HK. Safety of As-Needed Budesonide-Formoterol in Mild Asthma: Data from the Two Phase III SYGMA Studies. Drug Saf. 2021 Apr;44(4):467-478. doi: 10.1007/s40264-020-01041-z. Epub 2021 Feb 6. PMID 33548020
- [Derived] O'Byrne PM, FitzGerald JM, Bateman ED, Barnes PJ, Zheng J, Gustafson P, Lamarca R, Puu M, Keen C, Alagappan VKT, Reddel HK. Effect of a single day of increased as-needed budesonide-formoterol use on short-term risk of severe exacerbations in patients with mild asthma: a post-hoc analysis of the SYGMA 1 study. Lancet Respir Med. 2021 Feb;9(2):149-158. doi: 10.1016/S2213-2600(20)30416-1. Epub 2020 Oct 1. PMID 33010810
- [Derived] O'Byrne PM, FitzGerald JM, Bateman ED, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Ivanov S, Reddel HK. Inhaled Combined Budesonide-Formoterol as Needed in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1865-1876. doi: 10.1056/NEJMoa1715274. PMID 29768149
- [Derived] O'Byrne PM, FitzGerald JM, Zhong N, Bateman E, Barnes PJ, Keen C, Almqvist G, Pemberton K, Jorup C, Ivanov S, Reddel HK. The SYGMA programme of phase 3 trials to evaluate the efficacy and safety of budesonide/formoterol given 'as needed' in mild asthma: study protocols for two randomised controlled trials. Trials. 2017 Jan 10;18(1):12. doi: 10.1186/s13063-016-1731-4. PMID 28069068
- [Derived] Reddel HK, Busse WW, Pedersen S, Tan WC, Chen YZ, Jorup C, Lythgoe D, O'Byrne PM. Should recommendations about starting inhaled corticosteroid treatment for mild asthma be based on symptom frequency: a post-hoc efficacy analysis of the START study. Lancet. 2017 Jan 14;389(10065):157-166. doi: 10.1016/S0140-6736(16)31399-X. Epub 2016 Nov 30. PMID 27912982
- See also: D589SC00001-statistical-analysis-plan-edition-4_29Sep2017_pdfa — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2648&filename=D589SC00001-statistical-analysis-plan-edition-4_29Sep2017_pdfa.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5721 patients enrolled; 5003 run-in, 718 not run-in; 3849 randomised, 1154 not randomised: 1022 did not meet incl/excl criteria, 4 adverse event, 5 severe non-compliance to protocol, 104 subject decision, 7 subject lost to follow-up, 12 other reason.
Pre-assignment Details: Eligibility was assessed at Visits 1, 2, 3. IC obtained at V1. At V2, eligible patients stopped prescribed asthma medication and entered a 2-4 week run-in period, treated only with SABA Bricanyl Turbuhaler 0.5 mg, 'as needed'. Lung function was performed by spirometry to confirm eligibility. Eligible patients were randomised at Visit 3.
Groups:
- Placebo Bid + Symbicort 'as Needed': Placebo for budesonide (Placebo Turbuhaler) + Symbicort Turbuhaler (budesonide/formoterol 160/4.5 μg)
- Placebo Bid + Terbutaline 'as Needed': Placebo for budesonide (Placebo Turbuhaler) + Terbutaline Turbuhaler 0.4 mg 'as needed'
- Pulmicort Bid + Terbutaline 'as Needed': Pulmicort Turbuhaler (budesonide 200 μg) + Terbutaline Turbuhaler 0.4 mg 'as needed'
Period: Overall Study
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Started | 1277 | 1277 | 1282
Completed | 1144 | 1084 | 1135
Not Completed | 133 | 193 | 147
Not completed — Study specific withdrawal criteria | 4 | 21 | 6
Not completed — Other | 20 | 25 | 20
Not completed — Eligibility criteria not fulfilled | 9 | 14 | 8
Not completed — Withdrawal by Subject | 75 | 93 | 77
Not completed — Protocol Violation | 16 | 13 | 15
Not completed — Lost to Follow-up | 3 | 12 | 11
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 6 | 15 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set includes all patients randomised and receiving any IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed' | Total
Number analyzed (Participants) | 1277 | 1277 | 1282 | 3836
Age, Customized [Count of Participants; unit: Participants] — Age is being measured in years
  Participants
    >=12 - <18 | 161 | 144 | 173 | 478
    >=18 - <50 | 711 | 739 | 736 | 2186
    >=50 - <65 | 308 | 315 | 285 | 908
    >=65 - <85 | 97 | 78 | 87 | 262
    >=85 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 777 | 771 | 797 | 2345
  Male | 500 | 506 | 485 | 1491
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    American Indian Or Alaska Native | 74 | 73 | 73 | 220
    Asian | 340 | 336 | 347 | 1023
    Native Hawaiian Or Other Pacific Islander | 1 | 0 | 0 | 1
    Black Or African American | 24 | 33 | 24 | 81
    White | 721 | 726 | 728 | 2175
    Other | 117 | 109 | 110 | 336

OUTCOME MEASURES:

1. Primary Outcome: 'Well-controlled Asthma Week' - a Derived Binary Variable (Yes/No)
Description: A well-controlled asthma week is defined as the fulfilment of both conditions A) and B) below: A) Two or more of the following criteria are fulfilled: - No more than 2 days with a daily asthma symptom score >1 - No more than 2 days of 'as needed' medication use, up to a maximum of 4 occasions per week (multiple occasions per day should be regarded as separate occasions) - Morning PEF ≥80% of Predicted Normal every day B) Both of the following criteria are fulfilled: - No nighttime awakenings due to asthma - No additional inhaled and/or systemic glucocorticosteroid treatment due to asthma. The binary variable well-controlled asthma week was derived for each patient and study week. In addition, for each week, the percent of patients with well-controlled asthma week was derived. It is required that the eDiary had to be completed on at least 5 days in a week to be a well-controlled asthma week.
Time Frame: Weekly, up to 52 weeks
Population: Full analysis set. Patients with no evaluable weeks are not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Percentage | 34.4 (36.02) | 31.1 (34.90) | 44.4 (39.10)
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.046, Regression, Logistic; Repeated measures logistic regression, with treatment, pre-study treatment, region and study week as fixed effects; Odds Ratio (OR) = 1.14, 95% CI 2-sided [1.00 to 1.30] — An odds ratio greater than 1 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Non-Inferiority — Non-inferiority analysis based on CI instead of p-value, hence no p-value calculated for this analysis. Lower limit of the 2-sided 95% CI >=0.8 indicates Symbicort 'as needed' is non-inferior to Pulmicort bid; Regression, Logistic; Repeated measures logistic regression with treatment, pre-study treatment, region and study week as fixed effects; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.57 to 0.73]

2. Secondary Outcome: Number of Participants Experiencing at Least One Severe Asthma Exacerbation
Description: A severe exacerbation is defined as a deterioration of asthma requiring any of the following: use of systemic glucocorticosteroids (GCS) for at least 3 days, inpatient hospitalization, or emergency room visit due to asthma that required systemic steroids
Time Frame: Day 1 up to 52 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Participants | 71 | 152 | 78
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Regression, Cox; Cox-regression model with randomised treatment, pre-study treatment, severe exacerbations in the last 12 months (0, >=1) and region as covariates; Hazard Ratio (HR) = 0.435, 95% CI 2-sided [0.328 to 0.577] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first severe exacerbation
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.524, Regression, Cox; Cox regression model with randomised treatment, pre-study treatment, severe exacerbations in the last 12 months (0,>=1) and region as covariates; Hazard Ratio (HR) = 0.901, 95% CI 2-sided [0.653 to 1.242] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first severe exacerbation

3. Secondary Outcome: Number of Participants Experiencing at Least One Moderate or Severe Asthma Exacerbation
Description: A moderate exacerbation is defined as a deterioration of asthma requiring a change in treatment, i.e. initiation of prescribed additional ICS treatment to avoid progression of the worsening of asthma to a severe exacerbation.
  A severe exacerbation is defined as a deterioration of asthma requiring any of the following: use of systemic glucocorticosteroids (GCS) for at least 3 days, inpatient hospitalization, or emergency room visit due to asthma that required systemic steroids
Time Frame: Day 1 up to 52 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Participants | 131 | 274 | 143
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Regression, Cox; [statistical method as in outcome 2, analysis 2]; Hazard Ratio (HR) = 0.429, 95% CI 2-sided [0.348 to 0.528] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first moderate or severe exacerbation
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.436, Regression, Cox; [statistical method as in outcome 2, analysis 2]; Hazard Ratio (HR) = 0.910, 95% CI 2-sided [0.718 to 1.153] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Average Change From Baseline in Pre-dose Forced Expiratory Volume in 1 Second (FEV1)
Description: Overall estimate of FEV1 (mL) pre-bronchodilator change from baseline. Baseline is the measurement at Visit 3 (prior to first dose of Investigational Product) from MMRM (mixed model repeated measures analysis).
Time Frame: Study weeks 0,4,16,28,40,52
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
mL | 65 [47.6 to 82.4] | 11.2 [-6.4 to 28.9] | 119.3 [101.9 to 136.7]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; MMRM with treatment, pre-study treatment, region, visit and (treatment x visit) as fixed, patient as random and baseline FEV1 as continuous covariate; Mean Difference (Net) = 53.8, 95% CI 2-sided [29.1 to 78.5] — Mean difference greater than 0 favours Symbicort 'as needed'. This is the estimate across all treatment visits
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -54.3, 95% CI 2-sided [-78.8 to -29.8] — Mean difference greater than 0 favours Symbicort 'as needed'. This is the estimate across all treatment visits

5. Secondary Outcome: Average Change From Baseline in Morning Peak Expiratory Flow (PEF)
Description: Morning peak expiratory flow (eDiary) change from baseline over the randomised treatment period. Baseline is defined as the mean of all non-missing morning measurements during the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
L/min | -3.97 [-6.86 to -1.09] | -15.92 [-18.80 to -13.04] | 6.01 [3.13 to 8.88]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with randomised treatment, pre-study treatment and region as factors and baseline PEF as a continuous covariate; Mean Difference (Net) = 11.95, 95% CI 2-sided [7.89 to 16.00] — Mean difference greater than 0 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = -9.98, 95% CI 2-sided [-14.03 to -5.93] — Mean difference greater than 0 favours Symbicort 'as needed'

6. Secondary Outcome: Average Change From Baseline in Evening PEF
Description: Evening peak expiratory flow (eDiary) change from baseline during the randomised treatment period. Baseline is defined as the mean of all non-missing evening measurements during the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
L/min | -11.20 [-14.01 to -8.39] | -22.15 [-24.96 to -19.34] | -4.97 [-7.77 to -2.17]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = 10.94, 95% CI 2-sided [6.99 to 14.90] — Mean difference greater than 0 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.002, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = -6.23, 95% CI 2-sided [-10.18 to -2.29] — Mean difference greater than 0 favours Symbicort 'as needed'

7. Secondary Outcome: Average Change From Baseline in Number of Inhalations of 'as Needed' Medication.
Description: 'As needed' inhalations change from baseline over the randomised treatment period. Baseline is defined as the last 10 days of the run-in period. 'As needed' use was calculated as the cumulative doses of 'as needed' medication over the randomised treatment period divided by the follow-up time (number of days - 1). ie, average number of inhalations per day.
Time Frame: up to 52 weeks
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: Number of inhalations per day
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Number of inhalations per day | -0.95 (0.82) | -0.82 (0.92) | -1.06 (0.90)

8. Secondary Outcome: Average Change From Baseline in Asthma Symptom Score
Description: Asthma symptom score (eDiary) change from baseline during the randomised treatment period. Symptom score is entered morning and evening by the patient on a 4-point scale from 0 to 3 with higher values indicating more severe symptoms. Asthma symptom score is then the sum of the day and night scores, which implies a range of scores from 0 - 6, with higher values indicating more severe symptoms. Baseline is defined as the mean of all non-missing measurements during the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
units on a scale | -0.23 [-0.27 to -0.19] | -0.11 [-0.15 to -0.07] | -0.32 [-0.36 to -0.28]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model with randomised treatment, pre-study treatment and region as factors and baseline asthma symptom score as a continuous covariate; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.18 to -0.06] — Mean difference less than 0 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.004, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Net) = 0.09, 95% CI 2-sided [0.03 to 0.15] — Mean difference less than 0 favours Symbicort 'as needed'

9. Secondary Outcome: Change From Baseline in the Percentage of Nighttime Awakenings Due to Asthma
Description: Night-time awakenings (%) due to asthma change from baseline. Variable analysed is the proportion (%) of nights during the relevant period with night-time awakenings. Baseline refers to the last 10 nights of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: % of nights
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
% of nights | -7.5 (24.0) | -4.6 (23.4) | -9.8 (22.7)

10. Secondary Outcome: Change From Baseline in Percentage of Symptom-free Days
Description: Symptom-free days (%) change from baseline during the randomised treatment period.Variable analysed is the proportion (%) of symptom-free days during the relevant period. Baseline refers to the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
% of days | 4.2 (25.9) | 1.3 (24.8) | 6.8 (27.6)

11. Secondary Outcome: Change From Baseline in Percentage of 'As Needed' Free Days
Description: 'As needed' free days (%) change from baseline during the randomised treatment period. An 'as needed' free day is defined as a day and night with no use of 'as needed' medication. Variable analysed is the proportion (%) of 'as needed' free days during the relevant period. Baseline refers to the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
% of days | 44.2 (31.0) | 45.0 (30.7) | 51.7 (30.6)

12. Secondary Outcome: Change From Baseline in Percentage of Asthma Control Days
Description: Asthma control days (%) change from baseline. An asthma control day is defined as the fulfilment of all of the following criteria; a day and night with no asthma symptoms, a night with no awakenings due to asthma symptoms and a day and night with no use of 'as needed' medication. Variable analysed is the proportion (%) of asthma control days during the randomised treatment period. Baseline refers to the last 10 days of the run-in period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
% of days | 13.2 (23.9) | 12.8 (23.3) | 18.5 (28.4)

13. Secondary Outcome: Number of Patients With Study Specific Asthma Related Discontinuation
Description: Study specific asthma related discontinuation
Time Frame: up to 52 weeks
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Participants | 4 | 21 | 6

14. Secondary Outcome: Poorly Controlled Asthma Weeks
Description: A poorly-controlled asthma week is defined as a week meeting any one of the following conditions: Two or more consecutive days with awakenings due to asthma on both nights; A recorded use of 'as needed' medication for symptom relief of at least 3 occasions per day, for at least 2 consecutive days; Additional systemic GCS treatment required for severe exacerbation. If there were sufficient data within a week available to confirm the week was not poorly-controlled, the week is labelled as 'does not meet criteria for poorly-controlled'.
Time Frame: Weekly for up to 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
weeks | 7.7 (13.3) | 9.7 (13.8) | 6.7 (12.7)

15. Secondary Outcome: Number of Participants Experiencing at Least One Occasion With Additional Steroids for Asthma
Description: Additional steroids for asthma includes any additional inhaled and/or systemic glucocorticosteroids treatment due to asthma while in the randomised treatment period.
Time Frame: Day 1 up to 52 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
Participants | 164 | 345 | 187
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Regression, Cox; Cox regression model with randomised treatment, pre-study treatment and region as covariates; Hazard Ratio (HR) = 0.413, 95% CI 2-sided [0.343 to 0.497] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first additional steroids
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.175, Regression, Cox; Cox regression model with randomised treatment, pre-study treatment and region as covariates; Hazard Ratio (HR) = 0.865, 95% CI 2-sided [0.701 to 1.067] — A hazard ratio less than 1 indicates that Symbicort 'as needed' prolongs the time to first additional steroids

16. Secondary Outcome: Average Change From Baseline in Asthma Control Questionnaire (ACQ-5)
Description: Asthma Control Questionnaire 5-item version score change from baseline. ACQ questionnaire contains five questions on patients' symptoms, which are assessed on a 7-point scale from 0 (representing good control) to 6 (representing poor control). The score is the mean score of all questions for which responses are provided.
Time Frame: Study weeks 0,4,16,28,40,52
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
units on a scale | -0.33 [-0.36 to -0.29] | -0.17 [-0.21 to -0.14] | -0.48 [-0.51 to -0.44]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; MMRM with treatment, pre-study treatment, region, visit and (treatment x visit) as fixed, patient as random and baseline ACQ-5 as continuous covariate; Mean Difference (Net) = -0.154, 95% CI 2-sided [-0.203 to -0.105] — Mean difference less than 0 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = 0.149, 95% CI 2-sided [0.101 to 0.198] — Mean difference less than 0 favours Symbicort 'as needed'

17. Secondary Outcome: Average Change From Baseline in Asthma Quality of Life Questionnaire; Standard Version (AQLQ(S))
Description: Asthma Quality of Life Questionnaire Standardised Version (AQLQ (S) overall score change from baseline. AQLQ(S) consists of 32 questions in 4 domains. Each question is assessed on a 7-point scale from 1 to 7, with higher values indicating better health-related quality of life. The overall score is calculated as the mean score of all 32 items.
Time Frame: Study weeks 0,16,28,40,52
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
units on a scale | 0.313 [0.276 to 0.351] | 0.186 [0.148 to 0.225] | 0.415 [0.377 to 0.453]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; MMRM with treatment, pre-study treatment, region, visit and treatment x visit as fixed, patient as random and baseline AQLQ(S) as continuous covariate; Mean Difference (Net) = 0.127, 95% CI 2-sided [0.074 to 0.181] — Mean difference greater than 0 favours Symbicort 'as needed'
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 17, analysis 1]; Mean Difference (Net) = -0.102, 95% CI 2-sided [-0.155 to -0.049] — Mean difference greater than 0 favours Symbicort 'as needed'

18. Secondary Outcome: Percentage of Controller Use Days
Description: ICS controller use days (%) during the randomised treatment period is calculated as the cumulative number of days when any controller medication (containing ICS) was taken including maintenance (Pulmicort bid group) and 'as needed' medication (Symbicort 'as needed' group) and additional prescribed ICS for asthma exacerbations and/or long term poor asthma control (all treatment groups), divided by the number of days in the randomised treatment period.
Time Frame: up to 52 weeks
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: % of days
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
% of days | 30.8 (28.7) | 5.6 (16.8) | 85.6 (19.5)

19. Secondary Outcome: Annual Severe Asthma Exacerbation Rate
Description: Severe asthma exacerbations over the randomised treatment period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per year
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
exacerbations per year | 0.07 [0.06 to 0.09] | 0.20 [0.16 to 0.24] | 0.09 [0.07 to 0.11]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Negative binomial model; Negative binomial model with treatment, pre-study treatment, severe exacerbations in the last 12 months (0,>=1) and region as covariates; Rate ratio = 0.36, 95% CI 2-sided [0.27 to 0.49] — A rate ratio less than 1 indicates a lower rate of severe exacerbations in the Symbicort 'as needed' treatment group
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.279, Negative binomial model; [statistical method as in outcome 19, analysis 1]; Rate ratio = 0.83, 95% CI 2-sided [0.59 to 1.16] — A rate ratio less than 1 indicates a lower rate of severe exacerbations in the Symbicort 'as needed' treatment group

20. Secondary Outcome: Annual Moderate or Severe Asthma Exacerbation Rate
Description: Moderate or severe asthma exacerbations during the randomised treatment period.
Time Frame: up to 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per year
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
Number analyzed (Participants) | 1277 | 1277 | 1282
exacerbations per year | 0.14 [0.12 to 0.17] | 0.36 [0.31 to 0.42] | 0.15 [0.13 to 0.18]
Statistical Analysis 1: Comparison: Placebo Bid + Symbicort 'as Needed' vs Placebo Bid + Terbutaline 'as Needed'; Test type: Superiority; p < 0.001, Negative binomial model; [statistical method as in outcome 19, analysis 1]; Rate ratio = 0.40, 95% CI 2-sided [0.32 to 0.49] — A rate ratio less than 1 indicates a lower rate of moderate or severe exacerbations in the Symbicort 'as needed' treatment group
Statistical Analysis 2: Comparison: Placebo Bid + Symbicort 'as Needed' vs Pulmicort Bid + Terbutaline 'as Needed'; Test type: Superiority; p = 0.663, Negative binomial model; [statistical method as in outcome 19, analysis 1]; Rate ratio = 0.95, 95% CI 2-sided [0.74 to 1.21] — [estimate comment as in outcome 20, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were summarised from Visit 2 up to the follow-up visit at week 54. Serious adverse events were recorded from the time of informed consent up to the follow-up visit at week 54.
Arm/Group | Placebo Bid + Symbicort 'as Needed' | Placebo Bid + Terbutaline 'as Needed' | Pulmicort Bid + Terbutaline 'as Needed'
All-Cause Mortality (participants affected / at risk) | 0/1277 | 0/1277 | 2/1282
Serious Adverse Events (participants affected / at risk) | 38/1277 | 50/1277 | 37/1282
Other Adverse Events (participants affected / at risk) | 295/1277 | 378/1277 | 360/1282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Bid + Symbicort 'as Needed' (N=1277) | Placebo Bid + Terbutaline 'as Needed' (N=1277) | Pulmicort Bid + Terbutaline 'as Needed' (N=1282)
Abcess intestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atypical mycobacterial pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Keratitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leimyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 16 (22) | 8 (8)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chrondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolothiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lumbar limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patient-device incompatibility (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Bid + Symbicort 'as Needed' (N=1277) | Placebo Bid + Terbutaline 'as Needed' (N=1277) | Pulmicort Bid + Terbutaline 'as Needed' (N=1282)
Upper respiratory tract infection (Infections and infestations) | 71 (86) | 76 (95) | 93 (125)
Viral upper respiratory tract infection (Infections and infestations) | 75 (90) | 79 (95) | 84 (98)
Asthma (Respiratory, thoracic and mediastinal disorders) | 32 (40) | 95 (125) | 50 (61)
Pharyngitis (Infections and infestations) | 33 (39) | 34 (41) | 48 (54)
Bronchitis (Infections and infestations) | 33 (39) | 41 (44) | 37 (48)
Headache (Nervous system disorders) | 23 (44) | 25 (54) | 29 (32)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 28 (33) | 28 (32) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT02149199/SAP_000.pdf
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02149199/Prot_002.pdf